CLINICAL TRIAL: NCT04100954
Title: Cost-effectiveness Analysis of Vocal Rehabilitation With Strengthened Tracheoesophageal Voice Implant Prosthesis Versus Standard Voice Prosthesis in Case of Repeated Intra-prosthetic Leakage After Total Laryngectomy
Acronym: PHRASAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC19_0180
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Laryngectomy
Keywords: phonatory prosthesis; voice rehabilitation; reinforced voice prosthesis; laryngectomy; total pharyngolaryngectomy; total circular pharyngolaryngectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinforced prosthesis (Experimental): Implementation of a reinforced prosthesis with silver coating and double valve, whatever which type of prosthesis the patient previously had.
  Interventions: Device: Reinforced prosthesis
- Standard prosthesis (Active Comparator): Implementation of a standard prosthesis (simple valve, not reinforced), similar to the prosthesis the patient previously had.
  Interventions: Device: Standard prosthesis

INTERVENTIONS:
Device: Reinforced prosthesis — Implementation of a reinforced prosthesis during a medical consultation or under local anesthesia, after removal of the former prosthesis, in case of intraprothetic leakage.
  Arms: Reinforced prosthesis
Device: Standard prosthesis — Implementation of a standard prosthesis during a medical consultation or under local anesthesia, after removal of the former prosthesis, in case of intraprothetic leakage.
  Arms: Standard prosthesis

SUMMARY:
The purpose of this study is to determine the cost-effectiveness of vocal rehabilitation with reinforced inter-tracheoesophageal voice prosthesis versus standard voice prosthesis in case of repeated intra-prosthetic leakage in total laryngectomy patients.

This is a one year medico-economic study involving patients carrying a standard voice prosthesis implant and having undergone 2 successive prosthesis replacements within 3 months of interval and/or requiring at least 4 changes in the last 12 months, for intraprosthetic leakage.

Eligible subjects will be randomized in 2 groups: reinforced prosthesis with silver coating and double valve (Dual Valve) or standard prosthesis (single unreinforced valve), of the same model as the prosthesis previously implanted in the patient.

DETAILED DESCRIPTION:
Prosthetic voice rehabilitation is a widespread practice that allows the patient to resume phonation quickly after total laryngectomy/total pharyngolaryngectomy/total circular pharyngolaryngectomy.

When the longevity of the implant is abnormally short (less than 3 months), the multiplication of changes is likely to increase the risk of overall morbidity related to maintaining the functionality of the voice prosthesis and to alter the patient's quality of life.

Reinforced innovative prostheses, currently not supported by the French Social Security, delay the occurrence of intraprosthetic leakage compared to standard prostheses.

This study assesses the economic efficiency from a societal perspective and a one-year time horizon, from vocal rehabilitation with reinforced inter-tracheoesophageal prosthesis versus standard voice prosthesis in case of intra-tracheal leakage in total laryngectomy patients.

Patients are randomized in 2 arms. Arm A usual care with reinforced prosthesis, or arm B usual care with standard prosthesis. Each patient is followed during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated surgically by total laryngectomy or total pharyngolaryngectomy or total circular pharyngolaryngectomy and carrying a voice prosthesis for at least 12 months
* Patient carrying a standard voice prosthesis and having undergone 2 successive prosthesis replacements within 3 months of interval and/or requiring at least 4 changes in the last 12 months, for intraprosthetic leakage
* Patients carrying a voice prosthesis, irrespective of the mark/model, of diameters between 16 and 20 French, and of length between 6 and 14 mm.
* Prosthetic replacement available under local or general anaesthesia
* Patient with primary cancer remission status
* Patient agreeing to participate in the study and having given oral, express and informed consent

Exclusion Criteria:

* Patient with local, regional or metastatic tumor evolution
* Patient who has had a first voice prosthesis for less than 12 months.
* Patient with peri-prosthetic leakage
* Patient presenting a dysfunction of the voice prosthesis not linked to an intra-prosthetic leak
* Patients whose tracheal fistula is no longer opened, or justifying a new tracheoesophageal puncture
* Patients with a voice prosthesis of a diameter strictly greater than 20 French
* Patients with voice prosthesis of strictly less than 6 mm or greater than 14 mm length
* Patient under anti-fungal treatment during the month prior to inclusion
* Adult protected patients
* Inability to complete the questionnaires
* Patients with an estimated life expectancy of less than 1 year
* Patients not affiliated to French National Health care insurance
* Patients under the protection of Justice
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost-Effectiveness Ratio (cost per avoided prosthesis change), based on a societal perspective, comparing the use of a reinforced voice prosthesis to the use of a standard prosthesis | 12 months
  Effectiveness will be measured by the mean of number of prosthesis changes in each arm. Costs will be measured by 1) Outpatient resource consumption collected in a declarative patient questionnaire and 2) Hospital care resources using the database of the Medicalised Information System Program of each recruiting site

SECONDARY OUTCOMES:
Incremental cost-utility ratio, based on a societal perspective, comparing the use of a reinforced voice prosthesis to the use of a standard one | 12 months
  Utility will be measured by Quality Adjusted Life Year (QALYs) as estimated from responses to the Euroqol-5 Dimensions (EQ-5D 5L) health-related quality of life questionnaire. The questionnaire focuses on 5 dimensions: mobility, personal autonomy, current activities, pain/discomfort and anxiety/depression. For each of these dimensions, 5 answers are possible.
  Cost will be measured as described in the Primary Outome Measure
Quality of life using Euroqol-5 Dimensions (EQ-5D) questionnaire | Baseline, 3 months, 6 months, 9 months and 12 months and at each voice prosthesis replacement
  Score of EQ-5D 5L. health-related quality of life questionnaire. The questionnaire focuses on 5 dimensions: mobility, personal autonomy, current activities, pain/discomfort and anxiety/depression. For each of these dimensions, 5 answers are possible, each answer corresponds to a score ranging from 1 to 5.
Quality of life using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) | Baseline, at 3 months, 6 months, 9 months and 12 months
  Score of the QLQ-C30 questionnaire, including 30 questions assessing some aspects of the quality of life of cancer patients. The total score ranges from 0 to 100.
Quality of life using the Head and Neck Quality of Life Questionnaire (QLQ - H&N 35) | Baseline, 3 months, 6 months, 9 months and 12 months
  Score of the QLQ - H&N 35, including 35 questions assessing other aspects of quality of life in patients with head and neck cancer. The total score ranges from 0 to 100
Quality of voice | Baseline, 3 months, 6 months, 9 months and 12 months and at each voice prosthesis replacement
  score of the Voice Handicap Index: 10 items assessing the patient's voice, with 5 possible answers per item ranking from "never" to "always". The total score ranges from 0 to 120
Quality of voice assessed by the patient | Baseline, 3 months, 6 months, 9 months and 12 months
  Voice quality assessed by the patient and by a patient's relative with a numeric scale ranging from 0 "worst possible voice" to 10 "best possible voice", before and after each voice prosthesis change
Patient quality of voice assessed by the patient's relative | Baseline, at 3 months, 6 months, 9 months and 12 months
  Voice quality assessed by the patient's relative if present at time of prosthesis replacement, with a numeric scale ranging from 0 "worst possible voice" to 10 "best possible voice", before and after each voice prosthesis change
Trips induced by voice prosthesis replacement | 12 months
  Number of trips made by the patient for his prosthesis replacement, declared by the patient
Time spent out of home | 12 months
  Time spent by the patient out of home induced by voice prosthesis leaks, declared by the patient
Feeding interruption | 12 months
  Number of days or hours during which the patient could not eat due to voice prosthesis leak, declared by the patient
Interruption of oral communication | 12 months
  Number of days or hours during which the patient could not speak due to voice prosthesis leak, declared by the patient
Frequency of voice prosthesis replacements | 12 months
  Number of voice prosthesis replacements
Lifetime of voice prostheses | 12 months
  Date of voice prosthesis replacement
Complications due to voice prosthesis | 12 months
  Number and type of complications due to voice prosthesis
Patient's pain due to voice prosthesis replacement | at each prosthesis replacement, during the 12 months follow-up
  Pain due to voice prosthesis replacement assessed by a numeric scale ranging from 0 "no pain" to 10 "worst pain", asked to the patient before and after each voice prosthesis change
Patient's dysphagia due to voice prosthesis replacement | Baseline and at each prosthesis replacement
  Score of the Dysphagia Handicap Index 10 items assessing the patient's dysphagia, with 5 possible answers per item ranking from "never" to "always". Total score ranges from 0 to 120.
Annual net financial benefit of developping the use of reinforced prosthesis | 5 years
  Net financial benefit of the development of reinforced phonatory implants' compared to standard implants'use for patients treated with thyroid lobectomy and with repeated intraprosthetic dysfunction, through a Budget Impact Analysis (BIA) with a 5-years' time horizon and a National Health Insurance's perspective (NHI).
  Methods: Financial consequences for the NHI of several scenarii of development of the reinforced phonatory implants' will be represented in a table, year by year and over 5 years, in terms of cost per scenario and in terms of cost difference between the scenarii (showing savings or additional costs generated by choosing to develop the reinforced phonatory implant).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Malard, Md PhD, Principal Investigator — Nantes University Hospital
Locations (13):
- France (13):
  - Chu Bordeaux, Bordeaux
  - CHU CAEN, Caen
  - Chu Gui de Chauliac, Montpellier
  - Chu Nantes, Nantes
  - Chu Nimes, Nîmes
  - Clcc Institut Curie, Paris
  - Hopital Bichat, Paris
  - Hopital Tenon, Paris
  - Chru de Poitiers, Poitiers
  - Chru Pontchaillou, Rennes
  - Hopital Hautepierre, Strasbourg
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy